CLINICAL TRIAL: NCT00995241
Title: Pilot Study to Compare the Pharmacokinetics Parameters in Plasma and Intracellular of Raltegravir Administered Once a Day in Adult Patients Infected With HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAL-IC
Record Dates: First submitted 2009-10-07; First posted 2009-10-15 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: HIV Infections
Keywords: Raltegravir; intracellular concentration; plasmatic concentration; HIV; Treatment experienced
MeSH Terms: conditions — HIV Infections | interventions — Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Raltegravir 800 mg / 24 hours (Experimental): Raltegravir 800 mg / 24 hours
  Interventions: Drug: Raltegravir

INTERVENTIONS:
Drug: Raltegravir — Raltegravir 800 mg / 24 hours.
  Other Names: N/P

SUMMARY:
The purpose of this study is to compare plasma and intracellular pharmacokinetic parameters of raltegravir 800 mg administered once daily in HIV infected patients.

DETAILED DESCRIPTION:
HIV integrase is the enzyme responsible for transferring the DNA encoded by HIV to host chromosomes, a necessary step for the replication of retroviruses. Raltegravir (RAL) is the first integrase inhibitor approved for HIV treatment of patients infected by this virus. RAL has demonstrated a marked antiretroviral activity against HIV strains resistant to other antiretroviral drug families and high virological efficacy in patients pre-treated so as naïve to antiretroviral treatment. In addition, its safety profile is very favourable.

Unlike what happens with other antiretrovirals such as protease inhibitors, there is not a relationship between the virological response to antiretroviral treatment with RAL and the trough concentration of drug in plasma. Similarly, in vitro studies have shown that, after infection of cultured cells, the rate of viral replication measured by p24 antigen production was continuing inhibited even when RAL was washed from the culture medium from the 8 hours after infection, suggesting the possibility of a post-antibiotic effect of the drug. Either way, as in the case of transcriptase inhibitor nucleoside analogues, this lack of correlation between pharmacokinetics and pharmacodynamics of RAL may only be the result of intracellular accumulation of drug in blood lymphocytes peripheral, which in turn could be explained either by setting the RAL to the pre-integration complex or through the saturation of certain cellular transporters responsible for pumping the RAL from the inside out-cell (efflux transporters). Anyway, the result would be a greater RAL intracellular half-life than plasmatic, which would translate into a clinically persistent antiretroviral effect compared with its concentration in plasma.

Based on the above is possible to suggest that the average life of RAL was longer in the peripheral blood lymphocytes than in plasma, and that this intracellular increased half-life could explain the absence of relationship between trough RAL concentration and its virological efficacy, post-antibiotic effect of RAL found in some studies in vitro which, on the other hand, could be relevant to the possible once-daily administration of raltegravir.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. HIV documented infection.
3. Stable antiretroviral treatment for at least 4 weeks.
4. HIV viral load in plasma <50 copies / mL for at least 12 weeks
5. Voluntary written informed consent.

Exclusion Criteria:

1. AIDS-defining illness in the previous 4 weeks
2. Suspicion of inadequate adherence to antiretroviral therapy
3. In the case of women, pregnant or breastfeeding, or non-use of contraceptives
4. History or suspicion of failure to cooperate adequately
5. Concomitant therapy in the two weeks prior to inclusion in the study with atazanavir, tenofovir, NNRTI, rifampicin, inhibitors of proton pump or other drugs with known interactions with raltegravir.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Plasmatic and intracellular concentration of raltegravir | 10 days

SECONDARY OUTCOMES:
Clearance, CL/F | 10 days
Volume of distribution, V/F | 10 days
Elimination half-life, t1/2 | 10 days
Area under the plasma concentration-time curve during the dosing interval AUC0-24 | 10 days
Maximum concentration | 10 days
Time to maximum concentration, Tmax | 10 days
Minimum concentration | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Jose Molto, MD,PhD, Principal Investigator — Germans Trias i Pujol Hospital; Marta Valle, MD,PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona